CLINICAL TRIAL: NCT07225361
Title: Ublituximab (Briumvi) for Early Forms of Relapsing Multiple Sclerosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: TG Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Farrah Mateen, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00224712
Record Dates: First submitted 2025-10-29; First posted 2025-11-06 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis (MS) - Relapsing-remitting
Keywords: Ublituximab; Briumvi; Multiple Sclerosis; Relapsing Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — ublituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Participants with Relapsing Multiple Sclerosis (Experimental): Participants with Relapsing Multiple Sclerosis will be treated with Ublituximab for the duration of the study.
  Interventions: Drug: Ublituximab

INTERVENTIONS:
Drug: Ublituximab — Currently, many care plans may defer initiating high-efficacy DMTs, such as Ublituximab, for patients who previously would have been previously considered to have clinically isolated syndrome or not definite MS because of safety concerns. Recent label updates including a case of progressive multifocal leukoencephalopathy and transaminase elevations may exacerbate this worry. However, emerging evidence suggests treatment at the earliest timepoint has important, favourable impacts on long-term MS outcomes, far outweighing safety risks. Data in this early-diagnosis MS population are however lacking, and robust safety and tolerability data, underscored by biomarkers that are relevant to people with early MS, will guide prescribers in clinical decision making and likely encourage early MS treatment adoption.
  Other Names: Briumvi

SUMMARY:
In this prospective, open-label, single-arm, single-institution trial, the investigators will accomplish the following two aims:

1. study the safety and tolerability of Ublituximab (Briumvi) twice annually in participants with early MS over a treatment observation period of ~12 months.
2. study the pre- and post-treatment change in plasma neurofilament light chain, tested at baseline pre-Ublituximab treatment, and q24 weeks for 96 weeks post Ublituximab treatment initiation.

DETAILED DESCRIPTION:
PROCEDURES INVOLVED:

Participants will be enrolled for an estimated 96 weeks: Measurements will be requested every 24 weeks on a specifically designed survey instrument for participants. Participants will be asked to report medication dosing, adherence to medicine, tolerability, etc. as per Table 1. It is planned that each participant will be enrolled for 96 weeks (screening visit, baseline visit and four follow up visits at 24, 48, 72, and 96 weeks respectively) and would receive Ublituximab on an every 24 week schedule through regular clinical care. Notably, insurance may cover Ublituximab at an every 26 week schedule in which case accommodations will be made to have each study visit at q24-26 week intervals.

Participants will be contacted and interviewed every 24 weeks to ensure study procedures are going as planned, verify data reported on medication and MS disease history, and ensure study procedures are operating smoothly. Participants who do not complete the surveys within 7 days of the scheduled timing will be contacted by a study coordinator by phone up to 3 times. Participants will also be asked to report any medication changes, dose changes, or discontinuations if they occur at any point between study visits.

Participants will be enrolled until a total of 40 individual participants are reached. All scheduled events listed here will be part of the study and not part of routine clinical care. Study screening will continue until 40 participants are fully enrolled. Once 40 participants are enrolled, additional patients will not be screened or enrolled regardless of whether existing participants drop out of the study or are lost to follow-up. Five screen failures are estimated based on our study team's experience with ENHANCE (Ublituximab clinical trial). Once a participant is enrolled, the study will follow an intention to treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Meet 2024 Criteria for Multiple Sclerosis (Montalban et al.) as confirmed by a neurologist; Includes dissemination in space in two of five topographies (with optic nerve included) and/or biomarker evidence such as positive cerebrospinal fluid oligoclonal bands, elevated kappa free light chains, at least six central vein lesions, or at least one paramagnetic rim lesion;
* Adult age 18-70 years,
* EDSS <2.5,
* Able to provide individual informed consent,
* MRI brain available to confirm the diagnosis of MS with fewer than 10 demyelinating lesions,
* Diagnosis of MS within the past <5 years,
* Planning to start Ublituximab for the treatment of relapsing MS,

Exclusion Criteria:

* Prior exposure to Mavenclad, Lemtrada, Cyclophosphamide, stem cell transplant or related bone marrow suppressive treatment,
* Prior exposure to other B-cell depleting agent including Ocrelizumab, Rituximab, Ofatumumab, and Inebilizumab.
* Current clinical trial participant,
* Unable to speak a language for which translation can be found in the hospital system,
* Unclear documentation of MS diagnosis or prior or current MS treatment,
* Recent major surgical procedure in the past 6 months,
* History of life-threatening infusion reaction on Ublituximab or prior anti-CD20 therapy
* Active hepatitis B virus (HBV) confirmed by positive results for Hepatitis B surface antigen (HBsAg) and anti-HBV tests.
* Receipt of any live of live-attenuated vaccines within 4 weeks prior to first drug product administration
* Moribund status,
* Unable to provide consent voluntarily due to reasons of capacity or other reasons (e.g. incarcerated, etc.),
* Unwilling to undergo blood draws,
* Unable to access Ublituximab through clinical coverage throughout the full 96-week treatment study period,
* Unable to complete the study activities for any reason as deemed by the study investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2029-03-15 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in plasma neurofilament light chain | Time Frame: Baseline (pre-treatment), and at 24, 48, 72, and 96 weeks post-treatment initiation
  Change in plasma neurofilament light chain concentration from baseline (pre-Ublituximab IV) to follow-up visits while on treatment longitudinally.

SECONDARY OUTCOMES:
Safety of Ublituximab | From baseline through study completion, up to 96 weeks
  The severity as well as the number of adverse events (AEs) and serious adverse events (SAEs), laboratory abnormalities, and infusion-related reactions throughout the study period.

OTHER OUTCOMES:
Tolerability of Ublituximab | From baseline through study completion, up to 96 weeks.
  Number of participants that discontinue treatment or delay doses due to side effects, as assessed by participant self-report and clinician documentation.

CONTACTS AND LOCATIONS:
Overall Officials: Farrah J Mateen, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vermunt L, Otte M, Verberk IMW, Killestein J, Lemstra AW, van der Flier WM, Pijnenburg YAL, Vijverberg EGB, Bouwman FH, Gravesteijn G, van de Berg WDJ, Scheltens P, van Harten AC, Willemse EAJ, Teunissen CE. Age- and disease-specific reference values for neurofilament light presented in an online interactive support interface. Ann Clin Transl Neurol. 2022 Nov;9(11):1832-1837. doi: 10.1002/acn3.51676. Epub 2022 Oct 5. PMID 36196979
- [Background] Canto E, Barro C, Zhao C, Caillier SJ, Michalak Z, Bove R, Tomic D, Santaniello A, Haring DA, Hollenbach J, Henry RG, Cree BAC, Kappos L, Leppert D, Hauser SL, Benkert P, Oksenberg JR, Kuhle J. Association Between Serum Neurofilament Light Chain Levels and Long-term Disease Course Among Patients With Multiple Sclerosis Followed up for 12 Years. JAMA Neurol. 2019 Nov 1;76(11):1359-1366. doi: 10.1001/jamaneurol.2019.2137. PMID 31403661
- [Background] Fitzgerald KC, Sotirchos ES, Smith MD, Lord HN, DuVal A, Mowry EM, Calabresi PA. Contributors to Serum NfL Levels in People without Neurologic Disease. Ann Neurol. 2022 Oct;92(4):688-698. doi: 10.1002/ana.26446. Epub 2022 Jul 13. PMID 35730070
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Sotirchos ES, Fitzgerald KC, Singh CM, Smith MD, Reyes-Mantilla M, Hersh CM, Hyland MH, Canissario R, Simmons SB, Arrambide G, Montalban X, Comabella M, Naismith RT, Qiao M, Krupp LB, Nicholas JA, Akgun K, Ziemssen T, Rudick R, Fisher E, Bermel RA, Mowry EM, Calabresi PA. Associations of sNfL with clinico-radiological measures in a large MS population. Ann Clin Transl Neurol. 2023 Jan;10(1):84-97. doi: 10.1002/acn3.51704. Epub 2022 Nov 25. PMID 36427295
- [Background] Freedman MS, Abdelhak A, Bhutani MK, Freeman J, Gnanapavan S, Hussain S, Madiraju S, Paul F. The role of serum neurofilament light (sNfL) as a biomarker in multiple sclerosis: insights from a systematic review. J Neurol. 2025 May 15;272(6):400. doi: 10.1007/s00415-025-13093-1. PMID 40372550
- [Background] Steinman L, Fox E, Hartung HP, Alvarez E, Qian P, Wray S, Robertson D, Huang D, Selmaj K, Wynn D, Cutter G, Mok K, Hsu Y, Xu Y, Weiss MS, Bosco JA, Power SA, Lee L, Miskin HP, Cree BAC; ULTIMATE I and ULTIMATE II Investigators. Ublituximab versus Teriflunomide in Relapsing Multiple Sclerosis. N Engl J Med. 2022 Aug 25;387(8):704-714. doi: 10.1056/NEJMoa2201904. PMID 36001711
- [Background] Kanatas P, Stouras I, Stefanis L, Stathopoulos P. B-Cell-Directed Therapies: A New Era in Multiple Sclerosis Treatment. Can J Neurol Sci. 2023 May;50(3):355-364. doi: 10.1017/cjn.2022.60. Epub 2022 May 16. PMID 35570581